CLINICAL TRIAL: NCT04967924
Title: Effect of Sport Specific Training Versus Neuromuscular Training on Dynamic Balance, Mobility and Flexibility in Field Rugby Players With Non-specific Low Back Pain. A Randomized Clinical Trial
Brief Title: Sport Specific Training Versus Neuromuscular Training on Field Rugby Players.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0414 Maliah
Record Dates: First submitted 2021-07-19; First posted 2021-07-20 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Athletic Injuries
Keywords: dynamic balance, Low back pain, neuromuscular training
MeSH Terms: conditions — Athletic Injuries; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sports specific training (Experimental): Treatments will be provided in 30 mins per week for 3 consecutive weeks. Weight programs include closed chain exercises (squats, pushups) and open chain exercises (leg press, chest fly using dumbbell) Stretch shortening cycle (enhances performance through storage of elastic energy during eccentric phase and activation of stretch reflex).
  Interventions: Other: Sports specific training
- neuromuscular training (Active Comparator): Treatments will be provided in 30 mins per week for 3 consecutive weeks Proprioceptive Neuromuscular Facilitation (PNF)
  Interventions: Other: neuromuscular training

INTERVENTIONS:
Other: neuromuscular training — Treatments will be provided in 30 mins per week for 3 consecutive weeks Proprioceptive Neuromuscular Facilitation (PNF)
  Arms: neuromuscular training
Other: Sports specific training — Treatments will be provided in 30 mins per week for 3 consecutive weeks. Weight programs include closed chain exercises (squats, pushups) and open chain exercises (leg press, chest fly using dumbbell) Stretch shortening cycle (enhances performance through storage of elastic energy during eccentric phase and activation of stretch reflex).
  Arms: Sports specific training

SUMMARY:
Randomized Clinical Trial in rugby sports club in Lahore. A Sample size of 26 is calculated using epitol.Group A: Sports specific training Treatments will be provided in 30 mins per week for 3 consecutive weeks. Weight programs include closed chain exercises (squats, pushups) and open chain exercises (leg press, chest fly using dumbbell) Stretch shortening cycle (enhances performance through storage of elastic energy during eccentric phase and activation of stretch reflex).

Group B: neuromuscular training Treatments will be provided in 30 mins per week for 3 consecutive weeks Proprioceptive Neuromuscular Facilitation (PNF)

DETAILED DESCRIPTION:
Rugby require constant pace changes that generates high musculoskeletal demand in rugby one of the commonly affected area is low back pain that can affect player performance and can be accelerated by injury, health and lifestyle factors and possibly by joint pain or musculoskeletal disorders. Data will be collected from players in registered rugby clubs of district Lahore. Informed consents will be taken from all participants with the knowledge of aims and procedure. The results of this study will help to improve treatment protocols options for players how it affects the rehab process and how it affects the movement and pain how it affects the rehab process and how the pain restricts movements among rugby players. This study will be based on a randomized clinical trial used to study the different level of effectiveness of sports specific training versus neuromuscular training on dynamic balance mobility, flexibility in field rugby players. Subjects with low back pain meeting the predetermined inclusion & exclusion criteria will be divided into two groups by randomization to avoid any plagiarism. Dynamic Balance, measured with Star Excursion Balance Test; Active Range of Motion (ROM), using a manual goniometer and Lumbar Flexibility, assessed with Fingertip-to-floor test will be used for data collection. Subjects in one group will be treated with Bilateral stretches, contract-relax PNF stretching training and other will be treated with weight training, aerobic exercises. Each subject will receive a total four weeks treatment session, thirty minutes sessions will be performed once a week for three weeks. Three evaluations will be performed once before treatment One week after treatment and four week post treatment follow-ups. Sample size 26 each group contains 13 participants. All statistical analysis will be performed with spss16.0.

ELIGIBILITY:
Inclusion Criteria:

* Female rugby players
* Who had suffered minor musculoskeletal injuries that did not preclude their sports participation.
* Age ranges from 16-30
* Being able to cooperate

Exclusion Criteria:

* Players presenting injuries which implied radicular compromise (sciatic pain, etc.)
* Players who had suffered moderate or severe musculoskeletal injuries in the past 6 months which precluded their normal sports participation.
* Traumatic pain, fractures or ruptured ligaments.
* Inflammatory and Infectious conditions
* Any recent surgical intervention
* Tumors/malignancy of bone

Ages: 16 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2021-01-09 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Goniometer | 6 weeks
  To measure ROM at hip and knee joints
Star exclusion test | 6 weeks
  The test originally incorporated reaching in eight directions while standing on each foot. the 8 different directions are following: anterior, anteromedial, medial, posteromedial, posterior, posterolateral, lateral and anterolateral.
  SEBT performance scores using the following simple equations:
  Average distance in each direction (cm) = Reach 1 + Reach 2 + Reach 3 / 3
  Relative (normalised) distance in each direction (%) = Average distance in each direction / leg length * 100
Finger tip to floor test | 6 weeks
  The patient is asked to bend forward and attempt to reach for the floor with their fingertips. The physical therapist then measures the distance between the patient's right long finger and the floor using a standard measuring tape.
  Mean fingertip- to-floor test was 21.5 21.7cm (range, 0-48cm) for men and 19.6 22cm (range, 0-50cm) for women

SECONDARY OUTCOMES:
visual analogue scale for pain | 6 weeks
  Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, MS, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Espi-Lopez GV, Lopez-Martinez S, Ingles M, Serra-Ano P, Aguilar-Rodriguez M. Effect of manual therapy versus proprioceptive neuromuscular facilitation in dynamic balance, mobility and flexibility in field hockey players. A randomized controlled trial. Phys Ther Sport. 2018 Jul;32:173-179. doi: 10.1016/j.ptsp.2018.04.017. Epub 2018 Apr 22. PMID 29793126
- [Background] Filipa AR, Smith TR, Paterno MV, Ford KR, Hewett TE. Performance on the Star Excursion Balance Test predicts functional turnout angle in pre-pubescent female dancers. J Dance Med Sci. 2013 Dec;17(4):165-9. doi: 10.12678/1089-313x.17.4.165. PMID 24565332
- [Background] Amado-Bonilla E, Pintado-Vidal MI, Mangas-Borrego MI, Marchena-Ortiz E, Barrantes-Chacon J, Moran JM. Comment on "Reference Values of Total Lean Mass, Appendicular Lean Mass, and Fat Mass Measured with Dual-Energy X-ray Absorptiometry in a Healthy Mexican Population".https://www.ncbi.nlm.nih.gov/pubmed/27815567/. Calcif Tissue Int. 2017 Jun;100(6):653. doi: 10.1007/s00223-016-0204-9. Epub 2016 Nov 4. No abstract available.
- [Background] Wang L, Xiao Y, Tian T, Jin L, Lei Y, Finnell RH, Ren A. Corrigendum to "Digenic variants of planar cell polarity genes in human neural tube defect patients." Mol Genet Metab. 2018 May;124(1):94-100. doi:10.1016/j.ymgme.2018.03.005. Epub 2018 Mar 18. https://pubmed.ncbi.nlm.nih.gov/29573971/. Mol Genet Metab. 2021 Mar;132(3):211. doi: 10.1016/j.ymgme.2021.01.010. Epub 2021 Feb 10. No abstract available. PMID 33582009